CLINICAL TRIAL: NCT03596294
Title: A Single-center, Randomized, Double-blind, Two-period Cross-over Study to Investigate the Effect of Rifampicin on the Pharmacokinetics of Clazosentan in Healthy Male Subjects
Brief Title: A Study in Healthy Male Subjects to Investigate Whether Administration of Rifampicin Can Affect the Fate of Clazosentan in the Body of Clazosentan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-054-106; 2018-001607-36 (EudraCT Number)
Record Dates: First submitted 2018-07-05; First posted 2018-07-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — clazosentan; Rifampin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, two-period, cross-over Phase 1 study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence AB (Experimental): Period A:
  Saline + clazosentan
  Period B:
  Rifampicin + clazosentan
  Interventions: Drug: Clazosentan; Drug: Rifampicin; Other: Saline (0.9% sodium chloride)
- Treatment sequence BA (Experimental): Period B:
  Rifampicin + clazosentan
  Period A:
  Saline + clazosentan
  Interventions: Drug: Clazosentan; Drug: Rifampicin; Other: Saline (0.9% sodium chloride)

INTERVENTIONS:
Drug: Clazosentan — Continuous i.v. infusion of 15 mg/h of clazosentan for 3 h
Drug: Rifampicin — Single i.v. dose of 600 mg rifampicin for 30 min
Other: Saline (0.9% sodium chloride) — Single i.v infusion of 500 mL saline for 30 min

SUMMARY:
A study in healthy male subjects to investigate whether administration of rifampicin can affect the fate in the body (amount and time of presence in the blood) of clazosentan

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male subjects aged between 18 and 65 years (inclusive) at Screening.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at Screening.
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on the same arm, after 5 min in the supine position at Screening and on Day -1 of the first Period.
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

Study-specific criteria

- Acceptance for the duration of the study and for 3 months thereafter to use a condom and not to procreate.

Exclusion Criteria:

* Previous exposure to clazosentan.
* Previous exposure to rifampicin within 3 months prior to Screening.
* Known hypersensitivity to clazosentan or rifampicin or treatments of the same class, or any of their excipients.
* Known hypersensitivity or allergy to natural rubber latex.
* Participation in a clinical study involving study treatment administration within 3 months prior to Screening or in more than 4 clinical studies within 1 year prior to Screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
* Positive results for hepatitis B surface antigen or hepatitis C virus antibody at Screening.
* Positive results from the HIV serology at Screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
AUC from zero to time t of the last measured concentration above the limit of quantification | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles
AUC from zero to infinity (AUC0-inf) | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles
AUC from zero to 3 h (AUC0-3) | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles
The maximum plasma concentration (Cmax) | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles
Terminal half-life (t½) | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles
Total body clearance (CL) | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles
Volume of distribution at steady state (Vss) | 24 hours post treatment infusion initiation
  The plasma PK parameters of clazosentan will be derived by non-compartmental analysis of the plasma concentration-time profiles

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No